CLINICAL TRIAL: NCT04805905
Title: A Comparison of Skin Grafts Versus Local Flaps for Facial Skin Cancer From the Patient Perspective: A Feasibility Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Mark McRae, Principal Investigator, McMaster University
Other Study IDs: 8304
Record Dates: First submitted 2021-02-01; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Skin Cancer, Basal Cell; Skin Cancer; Skin Cancer, Non-Melanoma; Skin Cancers - Squamous Cell Carcinoma; Patient Satisfaction
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Skin graft
  Interventions: Other: FACE-Q patient reported outcome
- Local flap
  Interventions: Other: FACE-Q patient reported outcome

INTERVENTIONS:
Other: FACE-Q patient reported outcome — As both interventions of treatment are gold standards and clinical equipoise exists if one intervention is superior to the other, there is no true control group. However, for the purpose of the application, the local flap group will be chosen as the "control" group.
  Skin graft (Experimental): Participants in the experimental group will receive a skin graft and receive the FACE-Q skin cancer questionnaire pre- and post-treatment. There will also be photos taken of the patient's face along with the distributed questionnaires.
  Local flap (Control): Participants in the experimental group will receive a local flap and receive the FACE-Q questionnaire pre- and post-treatment.

SUMMARY:
A prospective single-centered feasibility study will be conducted. The purpose of the feasibility study is to define the variables to be included in a subsequent pilot study, assess the feasibility of conducting a prospective cohort study, and the logistics for the study (i.e., training, patient recruitment, data collection, statistical analysis, etc.).

DETAILED DESCRIPTION:
A prospective single-centered feasibility study will be conducted. The purpose of the feasibility study is to define the variables to be included in a subsequent pilot study, assess the feasibility of conducting a prospective cohort study, and the logistics for the study (i.e., training, patient recruitment, data collection, statistical analysis, etc.).

Upon completion of the feasibility study, a prospective pilot cohort study would be performed to measure outcomes using the FACE-Q Skin Cancer module for patients receiving skin grafting or local flaps after excision of facial skin cancers.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the study if:

* they are 18 years or older
* presenting for treatment of a suspected non-melanoma facial skin cancer, including pre-malignant cancers (i.e., actinic keratosis),
* and scheduled to undergo reconstruction with either a skin graft or local tissue flap.

Exclusion Criteria:

Patients will be excluded in the study if they:

* present with altered level of consciousness,
* cannot provide consent,
* have facial nerve injury/previous facial nerve injury, have Melanoma skin cancer or Merkel cell carcinoma based on pathology reports, have polytrauma/multiple injuries, are pregnant, are undergoing free flap reconstruction, have bone involvement, or if they are under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be included in the study if they are 18 years or older, presenting for treatment of a suspected non-melanoma facial skin cancer, including pre-malignant cancers (i.e., actinic keratosis), and scheduled to undergo reconstruction with either a skin graft or local tissue flap. Patients will be excluded in the study if they: present with altered level of consciousness, cannot provide consent, have facial nerve injury/previous facial nerve injury, have Melanoma skin cancer or Merkel cell carcinoma based on pathology reports, have polytrauma/multiple injuries, are pregnant, are undergoing free flap reconstruction, have bone involvement, or if they are under the age of 18.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 12 months
  Percent of patients who are recruited for the feasibility study
Retention rate | 3 months from surgery
  The number of patients who complete the secondary outcomes (FACE-Q scores) at 3 months
Compliance rate | 12 months
  Compliance rate of patients receiving a treatment and completing the expected treated
Eligible patients | 12 months
  Percent of patients who meet eligibility criteria for the feasibility study

SECONDARY OUTCOMES:
FACE-Q score | 12 months
  FACE-Q is a recently developed and validated patient reported outcome measure (PROM) tool that allows clinicians to assess patient perspectives after skin cancer surgery of the face.The PROM is used to assess the perspective and impact of skin cancer as well as its treatment on the patient's quality of life (QoL). Patients with skin cancer may have increased anxiety, social isolation, and cosmetic concerns after surgery. The FACE-Q utilizes five scales to measure the psychometric, QoL, patient experience, and cosmetic outcomes. Raw scores are transformed to a 0-100 scale with a higher score indicating a better outcome
Facial photos | 12 months
  Patient photos will be taken post-op at 2 weeks, 3 months, 6 months, and one-year post-operation, if feasible

IPD SHARING:
Plan to Share IPD: No